CLINICAL TRIAL: NCT03923725
Title: A Multi-centre Randomised Controlled Non-inferiority Trial to Compare the Efficacy, Safety and Tolerability of Triple Artemisinin-based Combination Therapies Versus First-line ACTs + Placebo for the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Africa
Brief Title: A Trial to Compare the Efficacy, Safety and Tolerability of Combinations of 3 Anti-malarial Drugs Against Combina-tions of 2 Anti-malarial Drugs.
Acronym: DeTACT-Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAL18004
Record Dates: First submitted 2019-04-09; First posted 2019-04-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Plasmodium Falciparum Malaria (Uncomplicated)
Keywords: Artemether; Lumefantrine; Amodiaquine; Artesunate; Piperaquine; Mefloquine; Triple Artemisinin-based Combination Therapy (TACT)
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Artemether-lumefantrine+amodiaquine (AL+AQ) (Experimental): Triple ACTs
  Interventions: Drug: Artemether-lumefantrine+ Amodiaquine (AL+AQ)
- artemether-lumefantrine+placebo (AL+PBO) (Active Comparator): ACTs
  Interventions: Drug: Artemether-lumefantrine + placebo (AL+PBO)
- Artesunate-mefloquine+Piperaquine (AS-MQ+PPQ) (Experimental): Triple ACTs
  Interventions: Drug: Artesunate-mefloquine+piperaquine (AS-MQ+PPQ)
- Artesunate-mefloquine+placebo (AS-MQ+PBO) (Active Comparator): ACTs
  Interventions: Drug: Artesunate-mefloquine+placebo (AS-MQ+PBO)

INTERVENTIONS:
Drug: Artemether-lumefantrine+ Amodiaquine (AL+AQ) — AL: Currently available as dispersible tablets containing 20 mg of artemether and 120 mg of lumefantrine, in a fixed-dose combination formulation. The flavoured dispersible tablet paediatric formulation facilitates use in young children.
  The dose of artemether-lumefantrine is administered approaching the WHO-recommended target ranges of artemether 5-24 mg/kg and lumefantrine 29-144 mg/kg over 3 days.
  AQ: is available as dispersible tablets of 40 mg. The weight-based treatment schedule aims for a dosage of approximately 10mg (4.5-15mg)/kg/day amodiaquine for three days.
  Arms: Artemether-lumefantrine+amodiaquine (AL+AQ)
Drug: Artemether-lumefantrine + placebo (AL+PBO) — AL: Currently available as dispersible tablets containing 20 mg of artemether and 120 mg of lumefantrine, in a fixed-dose combination formulation. The flavoured dispersible tablet paediatric formulation facilitates use in young children.
  The dose of artemether-lumefantrine is administered approaching the WHO-recommended target ranges of artemether 5-24 mg/kg and lumefantrine 29-144 mg/kg over 3 days.
  PBO: Placebo tablets for amodiaquine are identical in size, shape and color to the amodiaquine tablets.
  Arms: artemether-lumefantrine+placebo (AL+PBO)
Drug: Artesunate-mefloquine+piperaquine (AS-MQ+PPQ) — AS: Artesunate will be administered according to an optimised dosing schedule using tablets of 32 or 100 mg artesunate with a dosing target of 4 mg/kg/day.
  MQ: Mefloquine will be administered according to an optimised dosing schedule using tablets of 70 or 220 mg mefloquine hydrochloride with a dosing target of 8.3 mg/kg/day.
  PPQ: Piperaquine will be administered according to an optimised dosing schedule using tablets of 160 or 500 mg of piperaquine tetraphosphate. The weight-based treatment aims for a dosage of approximately.
  * 24 mg/kg/day in patients <25 kg (range 16.0 - 32.0 mg/kg) piperaquine for three days, thereby approaching the WHO-recommended target range of 20 - 32 mg/kg per day.
  * 18 mg/kg/day in patients ≥25 kg (range 15.0 - 29.4 mg/kg) piperaquine for three days, thereby approaching the WHO-recommended target range of 16 - 27 mg/kg per day.
  Arms: Artesunate-mefloquine+Piperaquine (AS-MQ+PPQ)
Drug: Artesunate-mefloquine+placebo (AS-MQ+PBO) — AS: Artesunate will be administered according to an optimised dosing schedule using tablets of 32 or 100 mg artesunate with a dosing target of 4 mg/kg/day.
  MQ: Mefloquine will be administered according to an optimised dosing schedule using tablets of 70 or 220 mg mefloquine hydrochloride with a dosing target of 8.3 mg/kg/day.
  PBO: Placebo tablets for piperaquine are identical in size, shape and colour to the piperaquine tablets.
  Arms: Artesunate-mefloquine+placebo (AS-MQ+PBO)

SUMMARY:
A partially blinded randomised controlled non-inferiority trial comparing the efficacy, tolerability and safety of Triple ACTs artemether-lumefantrine+amodiaquine (AL+AQ) and artesunate-mefloquine+piperaquine (ASMQ+PPQ) and the ACTs artemether-lumefantrine+placebo (AL+PBO), artesunate-mefloquine+placebo (ASMQ+PBO) (with single-low dose primaquine in some sites) for the treatment of uncomplicated Plasmodium falciparum malaria to assess and compare their efficacy, safety, tolerability.

DETAILED DESCRIPTION:
Subjects will be randomized to up to four arms: artemether-lumefantrine + amodiaquine, artemether-lumefantrine + placebo, artesunate-mefloquine + piperaquine and artesunate-mefloquine + placebo. As a contingency measure in case of significant differences in the efficacy or safety of one of the combinations being tested and/or study drug expiry or unavailability, subjects may be randomised to 2 arms with a matching ACT-TACT pair, i.e., with artemether-lumefantrine + placebo or artemether-lumefantrine + amodiaquine OR artesunate-mefloquine + placebo or artesunate-mefloquine + piperaquine.

Some sites may randomize between 2 arms only with matching ACT-TACT pairs, i.e., artemether-lumefantrine + placebo or artemether-lumefantrine + amodiaquine OR artesunate-mefloquine + placebo or artesunate-mefloquine + piperaquine. In Rwanda, subjects will be randomized between 2 arms consisting of artemether-lumefantrine + placebo or artemether-lumefantrine + amodiaquine.

In the control arms, the ACT will be co-packed with a matched (appearance) placebo.

In lower transmission settings (Annual Parasite Incidence <50 per 1000 population per year) the treatment will include a single 0.25 mg/kg gametocytocidal dose of primaquine as recommended by the WHO for children ≥10 kg. All drug administrations will be observed.

Subjects will be treated in an in-patient unit for 3 days and followed up weekly up to D63. Microscopy to detect and quantify malaria parasitaemia will be performed daily (more frequently in patients with parasite density of >5000/µL at inclusion) during hospitalization, at all weekly and unscheduled visits. A physical examination and measurements of vital signs along with a symptom questionnaire for tolerability will be performed and recorded through a standardized method at baseline, daily during admission and weekly during follow up through D42 and at all unscheduled visits. Physical exam, vital sign measurements and assessments of symptoms will be performed on D49, D56, and D63 only for patients who are parasitaemic or those who report fever or other symptoms. Electrocardiographs will be performed during admission (H0, H4, H52 or H64) and day 42 of follow up to assess and compare the effect of ACTs and TACTs antimalarials on QT or QTc intervals.

The DeTACT-Africa Trial is funded by UK Aid from the UK government's Foreign, Commonwealth and Development Office.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥6 months to <12 years (For Gambia, Rwanda sites only: ≥6 months)
* Ability to take oral medication
* Acute uncomplicated P. falciparum monoinfection
* Asexual P. falciparum parasitaemia: 1,000/µL to ≤10% parasitaemia, determined on a peripheral blood film (At Gambia, Rwanda sites only: For subjects ≥12 years - 1000/µL to 200,000/µL)
* Fever defined as ≥ 37.5°C tympanic temperature or a history of fever within the last 24 hours
* Written informed consent by the subject or by parent/guardian in case of children lower than the age of consent and assent if required (per local regulations)
* Willingness and ability of the subjects or parents/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe malaria (adapted from WHO criteria)
* Patients not fulfilling criteria for severe malaria but with another indication for parenteral antimalarial treatment at the discretion of the treating physician
* Haematocrit <15% at screening (For Gambia, Rwanda sites only: For subjects ≥12 years - Haematocrit <20% at screening)
* Subjects who have received artemisinin or a derivative within the previous 7 days OR lumefantrine or amodiaquine within the previous 14 days OR mefloquine or piperaquine within the previous 30 days
* In applicable countries: use of seasonal malaria chemoprophylaxis (SMC) within the last 14 days.
* Acute illness other than malaria requiring systemic treatment
* Severe acute malnutrition (in Niger only - only those patients with Severe Acute Malnutrition and complications requiring inpatient nutritional treatment will be excluded)
* Known HIV infection
* Known tuberculosis infection
* For females: post-menarche (For Gambia, Rwanda sites only: females who are pregnant, trying to get pregnant or are lactating)
* History of allergy or known contraindication to any of the study drugs, including neuropsychiatric disorders and epilepsy
* Previous splenectomy
* Enrolment in DeTACT in the previous 3 months
* Participation in another interventional study in the previous 3 months

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2583 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
42 days Efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR). | 42 days
  42 days Efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR).

SECONDARY OUTCOMES:
63-day PCR corrected and uncorrected efficacy | 63 days
42-day PCR uncorrected efficacy | 42 days
Parasite clearance half-life | 3 Days
  Assessed by microscopy as primary parameter to determine parasite clearance
Proportion of subjects with microscopically detectable P. falciparum parasitaemia | Day 3
Fever clearance time | 63 Days
  fever clearance time (i.e. the time taken for the tympanic temperature to fall below 37.5 ºC)
Proportion of subjects with gametocytaemia | 63 Days
  proportion of subjects with gametocytaemia during and after treatment stratified by presence of gametocytes at enrolment
Incidence of adverse events | 42 days
  including markers of hepatic, renal or bone marrow toxicity; cardiotoxicity
Incidence of serious adverse events | 42 days
  including markers of hepatic, renal or bone marrow toxicity; cardiotoxicity
Number of cardiotoxicity events | 52 or 64 hours depends on treatment arm
  In particular QT or QTc-interval above 500 ms at timepoint H4 and H52/H64 and between these time points
Change in haemoglobin stratified for G6PD status/genotype | 28 days
Proportion of subjects requiring retreatment due to vomiting | 1 hour
  Proportion of subjects requiring retreatment due to vomiting within 1 hour after administration of the study drugs
Proportion of subjects that reports completing a full course of observed TACT | 3 days
Proportion of subjects that reports completing a full course of observed ACT | 3 days
proportion of subjects that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study because of drug related serious adverse event. | 42 days
Pharmacokinetic profiles | 42 days
  including Cmax and AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated subjects in correlation with pharmacodynamics measures of drug efficacy
Pharmacokinetic interactions | 42 days
  including Cmax and AUC) of artemisinin-derivatives and partner drugs in ACT and TACT treated subjects in correlation with pharmacodynamics measures of drug efficacy
Plasma levels of partner drugs | 7 days
  Plasma levels of partner drugs in correlation with treatment efficacy and treatment arm

OTHER OUTCOMES:
Comparison of 63-day vs 42-day PCR corrected and uncorrected efficacy | 63 days
  Comparison of 63-day vs 42-day PCR corrected and uncorrected efficacy of ACTs vs TACTs
Proportions of recurrent infections | 63 days
  Proportions of recurrent infections with parasites carrying mutations of known functional significance
Proportions of specimens collected at baseline with parasites carrying mutations | baseline
  Proportions of specimens collected at baseline with parasites carrying mutations of known functional or operational significance (pfkelch13, pfcrt, pfmdr1, pfdhfr, pfdhps, pfplasmepsin2 , partial or complete deletions of pfhrp2 and other current parasite genetic markers associated with resistance or identified over the course of the study)
Candidate markers of resistance | 63 days
  Candidate markers of resistance identified through genome wide association studies with in vivo or in vitro parasite drug sensitivity phenotypes
In vitro sensitivity of P. falciparum to artemisinins and partner drugs | 63 days.
  In vitro sensitivity of P. falciparum to artemisinins and partner drugs according to study sites and genotype
Accuracy of SNPs assessment | 63 days.
  Accuracy of SNPs assessment from dry blood spots versus from whole genome sequencing in leukocyte depleted blood samples
Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics | 14 days
Correlation of parasite clearance metrics as assessed by microscopy versus digital microscopy | 3 days
Comparison of transcriptomic patterns of drug sensitive and resistant parasites | 63 days
  Comparison of transcriptomic patterns of drug sensitive and resistant parasites before treatment and 6, 12 and 24 hours after start of treatment
Levels of RNA transcription coding for male or female specific gametocytes | 14 days
  Levels of RNA transcription coding for male or female specific gametocytes at admission up to day 14, stratified by the presence of gametocytes at enrolment
Correlation between the host genotype and the pharmacokinetics and pharmacodynamics of antimalarials. | 42 days
  Host genotype (e.g., CYP2D6, CYP3A4, KCNQ1/LQT1, KCNH2/LQT2, SCN5A/LQT3)
Correlations between the place of residence, work, recent travel history | 63 days
  Correlations between the place of residence, work, recent travel history assessed by interview and mobile phone records to identify behaviours and risk factors associated with malaria infection.
Correlation between titres of antibodies against malaria parasite antigens and - efficacy defined as PCR corrected adequate clinical and parasitological response (ACPR) - efficacy defined as adequate clinical and parasitological response (ACPR) | 63 days

CONTACTS AND LOCATIONS:
Locations (8):
- Institut des Sciences et Techniques (INSTech), Bobo-Dioulasso, Burkina Faso
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Centre National de Formation et de Recherche en Santé Rurale de Mafèrinyah, Conakry, Guinea
- Centre for Malaria and Other Tropical Diseases (CEMTROD), Ilorin, Kwara State, Nigeria
- Epicentre Niger, Niamey, Niger
- College of Medicine and Health Sciences, University of Rwanda, Kigali, Rwanda
- National Institute For Medical Research (NIMR), Tanga Medical Research Centre, Tanga, Tanzania
- MRC Unit The Gambia at LSHTM, Fajara, City of Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with data repositories such as the WorldWide Antimalarial Resistance Network (WWARN, terms of submission here: http://www.wwarn.org/tools-resources/terms-submission) or other researchers to use in the future. All personal information will be anonymised so that no individual can be identified from their treatment records, through interviews, or from mapping data.
Time Frame: After completion of trial activities and reporting.
Access Criteria: MORU Data Sharing Policy https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing WWARN Terms of Data Access https://www.wwarn.org/tools-resources/terms-data-access

DOCUMENTS (2):
  • Study Protocol (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03923725/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/25/NCT03923725/SAP_003.pdf